CLINICAL TRIAL: NCT07253558
Title: Effects of Music-Based Occupational Therapy Activities on Attention and Executive Functions in Children With Attention Deficit and Hyperactivity Disorder
Brief Title: Effects of Music-Based Occupational Therapy on Attention and Executive Functions in Children With ADHD
Acronym: MBOT-ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Principal Investigator, Ibrahim Erarslan, Principal Investigator and Research Assistant, Department of Occupational Therapy, Istanbul Medipol University; PhD Student, Health Sciences University, Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-2028
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Attention Deficit and Hyperactivity Disorder (ADHD)
Keywords: ADHD; Attention; Caregiver; Executive functions; Music-based activities
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The study was based on an occupational therapy-centered intervention model designed to enhance attention and executive functioning skills in children with attention deficit hyperactivity disorder (ADHD). The intervention model consisted of two structured therapeutic approaches. The first, the Occupational Therapy-Based Music Activity Model, integrated core principles of sensory integration, motor planning, and emotional regulation through rhythmic and interactive musical experiences. This approach emphasized active engagement, auditory-motor coordination, and task-oriented participation, aiming to support sustained attention, impulse control, and goal-directed behavior. The music-based sessions were delivered by an occupational therapist using structured group activities involving rhythm instruments, body movements, and attention-focused musical games.
  The second model, the Structured Occupational Therapy ADHD Protocol, served as the control intervention and was developed in accordance
Masking Description: Not applicable. This is an open-label single-arm study. The intervention was openly delivered to all participants by the same occupational therapist. No blinding was applied to participants or outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music-Based Occupational Therapy (Experimental): Participants in the experimental group received music-based occupational therapy for children with ADHD. The sessions were held once a week for six weeks, each lasting approximately 45 minutes. During the sessions, occupational therapy-based music activities were conducted using harmonicas and drums. These instruments were selected for their therapeutic potential to enhance fine motor skills, provide oral-motor sensory input, and promote rhythmic coordination. Sessions were conducted individually in a clinical environment and aimed to improve attention, executive functions, and caregiver-related outcomes.
  Interventions: Behavioral: Music-Based Occupational Therapy

INTERVENTIONS:
Behavioral: Music-Based Occupational Therapy — This behavioral intervention consisted of six weeks of occupational therapy-based music sessions lasting 45 minutes each, performed once a week. The intervention involved therapeutic use of harmonica and drums integrated into occupational therapy sessions to support sensory processing, attention, and motor planning in children with ADHD. The approach focused on enhancing attention, executive function, play skills, and self-regulation through rhythm-based sensory and motor engagement.

SUMMARY:
Attention Deficit/Hyperactivity Disorder (ADHD) is a neurodevelopmental condition that affects children's attention, behavior, and emotional regulation. This study examined whether occupational therapy sessions that include structured music activities can improve attention and executive functions in children with ADHD compared to standard occupational therapy. Thirty-nine children aged 6 to 17 participated and were randomly assigned to two groups. The music-based group received 45-minute sessions once a week for six weeks using harmonica and drum activities, while the control group received standard occupational therapy. Children's attention, executive skills, and caregiver stress were measured before and after the intervention using standardized parent-report scales. Both groups improved after therapy, but the music-based occupational therapy group showed greater gains in attention.

DETAILED DESCRIPTION:
Attention Deficit/Hyperactivity Disorder (ADHD) is a complex neurodevelopmental condition that affects attention, motor control, and executive functioning. In addition to pharmacological approaches, behavioral and sensory-based occupational therapy interventions are increasingly being used to support self-regulation and participation in daily activities.

This randomized controlled study was conducted to evaluate the effects of occupational therapy-based music activities on attention, executive functions, and caregiver burden in children with ADHD. Thirty-nine children aged 6-17 years with a clinical diagnosis of ADHD were included. Participants were randomly assigned to the experimental group (occupational therapy-based music; n=19) or the control group (standard occupational therapy; n=20). The intervention group received 45-minute sessions once a week for six consecutive weeks. The sessions incorporated harmonica and drum activities to enhance rhythmic coordination, sensory processing, and cognitive engagement within the occupational therapy framework. The control group received standard occupational therapy during the same period, focusing on activity organization, attention training, and behavioral strategies. Outcome measures were collected at baseline and at the end of the sixth week. Attention was assessed with the DSM-V Level 2 Inattention Scale, executive functions with the Childhood Executive Function Inventory (CHEXI), and caregiver burden with the Zarit Caregiver Burden Scale. Statistical analyses revealed significant improvements in all variables in both groups, with a greater effect on attention levels in the music-based occupational therapy group. These findings suggest that structured music-based occupational therapy can be an effective complementary intervention to improve attention, executive function, and family well-being in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ADHD
* Being between 5 and 12 years of age.
* Residing in Istanbul.
* The caregiver scoring 21 or above on the Parental Stress Index (PSI).
* The caregiver being between 18 and 65 years of age

Exclusion Criteria:

* Having an additional diagnosis accompanying ADHD.
* Having experienced a cardiopulmonary problem within the last 3 months.
* Having previously learned to play a musical instrument.
* The caregiver scoring 31 or above on the Beck Depression Inventory (BDI).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Attention Performance | Baseline and 6 weeks after intervention.
  Change in attention performance of children with ADHD after six weeks of music-based occupational therapy. Attention levels are assessed using the DSM-V Level 2 Inattention Scale, an 8-item parent-report questionnaire that evaluates inattention symptoms during the past seven days. The DSM-5 Level 2 Inattention Scale provides a four-point Likert-type assessment for screening inattention (0 = none, 1 = a little, 2 = quite a bit, 3 = very much). The sum of the scores obtained from the eight items can range between 0 and 24. A higher score indicates greater severity of inattention.

SECONDARY OUTCOMES:
Executive Function Skills | Baseline and 6 weeks after intervention.
  Change in executive function skills, including working memory, inhibition, planning, and regulation, after six weeks of music-based occupational therapy. Executive functions are assessed using the Childhood Executive Functioning Inventory (CHEXI) - Parent Form. The CHEXI (Childhood Executive Function Inventory), which consists of 26 items, is divided into four subscales: working memory (9 items), planning (6 items), inhibition (6 items), and regulation (5 items). The questions are answered by either parents or teachers. Each item uses a 1-to-5 scale to rate the degree of accuracy of the statement (1: absolutely not true, 5: absolutely true). The parent is asked to indicate how well the child fits that statement by selecting the appropriate number. As the total score obtained from the CHEXI increases, the child's executive functions weaken.
Caregiver Burden Level | Baseline and 6 weeks after intervention.
  Change in caregiver burden levels after the six-week music-based occupational therapy program. Caregiver burden is assessed using the Zarit Burden Interview (ZBI), which measures the physical, emotional, and social impact of care responsibilities on the primary caregiver. The total score of the scale ranges between 19 and 95, and the higher the score, the higher the burden experienced by the individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical considerations and privacy protection of child participants. The data include sensitive clinical and psychological information that cannot be anonymized sufficiently for open sharing. Only aggregated results will be reported in publications.

REFERENCES:
- [Background] Yeniceli D, Sener E, Korkmaz OT, Dogrukol-Ak D, Tuncel N. A simple and sensitive LC-ESI-MS (ion trap) method for the determination of bupropion and its major metabolite, hydroxybupropion in rat plasma and brain microdialysates. Talanta. 2011 Mar 15;84(1):19-26. doi: 10.1016/j.talanta.2010.11.063. Epub 2010 Dec 21. PMID 21315892
- See also: Case report published in Cureus related to therapeutic interventions in ADHD (PDF). — https://assets.cureus.com/uploads/case_report/pdf/260461/20240725-319105-fnbtv7.pdf
- See also: Research article published in DergiPark related to occupational therapy-based interventions in children with ADHD. — https://dergipark.org.tr/en/download/article-file/3750541

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT07253558/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT07253558/ICF_001.pdf